CLINICAL TRIAL: NCT01368705
Title: Determination of Protein Needs Using Nitrogen Balance in Infants Immediately Post Cardiothoracic Surgery
Brief Title: Nitrogen Balance in Infants After Post Cardiothoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Emeritus Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000012920
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Congenital Heart Disease
Keywords: Infants; Nitrogen Balance; Cardiothoracic surgery; Congenital heart disease; Malnutrition
MeSH Terms: conditions — Heart Defects, Congenital; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Active Comparator)
  Interventions: Dietary Supplement: Standard protein delivery
- Intervention Group 1 (Experimental)
  Interventions: Dietary Supplement: Intervention 1 (2.2g/kg/day)
- Intervention Group 2 (Experimental)
  Interventions: Dietary Supplement: Intervention 2 (3.0 g/kg/day)

INTERVENTIONS:
Dietary Supplement: Standard protein delivery — Protein delivery of 1.5 g/kg/day.
  Arms: Control Group
Dietary Supplement: Intervention 1 (2.2g/kg/day) — protein delivery of 2.2g/kg/day
  Arms: Intervention Group 1
Dietary Supplement: Intervention 2 (3.0 g/kg/day) — protein delivery of 3.0 g/kg/day
  Arms: Intervention Group 2

SUMMARY:
The objective is to the amount of protein infants require after cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
Postoperative neonates are susceptible to the adverse effects of surgery that is characterized by a breakdown of body stores. Without appropriate nutritional consideration this process can lead to increased physiological instability. It has been extensively documented that critically ill patients are typically catabolic. This results in body nitrogen losses from the breakdown of somatic protein to fuel metabolic processes such as, gluconeogenesis. The evaluation of this catabolic response is particularly crucial in infants due to their limited fat and lean body mass reserves. Quantifying the amount of protein needed to maintain body composition and to meet the demands of surgical stress is of clinical importance when considering factors associated with postoperative morbidity, such as delayed wound healing, impaired growth and prolonged hospital stay.

The results obtained from this study will assist with determining an appropriate level of protein for the development of optimal nutrition prescriptions that are aimed at reducing catabolism of body stores.

ELIGIBILITY:
Inclusion Criteria:

* Clinical decision to initiate parenteral nutrition based on determination by medical team
* Gestational age ≥ 35 weeks
* Birth weight ≥ 2000 grams
* Indwelling urinary catheters for urine collection
* Central venous access for parenteral nutrition

Exclusion Criteria:

* Chromosomal abnormalities known to effect protein metabolism
* Hepatic failure defined as ALT and AST > 500 UL with an INR > 2.5, not accounted for by therapeutic anticoagulation
* Renal failure defined as creatinine 2x the upper limit of normal for age.
* Sepsis or suspected sepsis, defined as clinical suspicion or confirmation of a systemic infection treated with antibiotics
* Excessive blood loss from chest tubes (5 ml/kg/hr) that has not resolved within six hours following admission to the CCCU; as indicated by the need for frequent blood transfusion these subjects will be withdrawn from the study
* Requiring Extra Corporeal Membrane Oxygenation (ECMO) support

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Nitrogen Balance | From 0-84 hours
  After an initial adaptation period of approximately 12 hours receiving parenteral nutrition the first 24-hour urine collection for nitrogen balance will be started; following this two successive 24-hour urine collections will be performed in order to obtain a three-day collection for nitrogen balance analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Pencharz, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada